CLINICAL TRIAL: NCT00048087
Title: A Phase II Study of ZD1839 (Iressa), Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor, in Combination With Docetaxel in Patients With Recurrent or Metastatic Advanced Non-Small Cell Lung Cancer
Brief Title: Iressa/Docetaxel in Non-Small-Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AstraZeneca (Industry); Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-004
Record Dates: First submitted 2002-10-24; First posted 2002-10-25 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Iressa + Docetaxel (Experimental)
  Interventions: Drug: ZD1839; Drug: Docetaxel

INTERVENTIONS:
Drug: ZD1839 — 250 mg by mouth daily each day for 4 weeks.
  Other Names: Iressa; Gefitinib
Drug: Docetaxel — 30 mg/m2 by IV on day 1 weekly for the first 3 weeks of each 4 week course.
  Other Names: Taxotere

SUMMARY:
Patients will receive 250 mg Iressa by mouth daily each day while on this study. Patients will also receive docetaxel 30 mg/m2 by by vein (IV) on day 1 weekly for the first 3 weeks of each course of therapy. A course of therapy is 4 weeks. Patients will not receive docetaxel during week 4. A maximum of 8 full cycles of docetaxel plus Iressa are planned. Patients may continue on daily Iressa until progressive disease and/or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed non-small cell lung cancer.
* Measurable, evaluable disease outside of a radiation port.
* ECOG performance status 0-2.
* Adequate hematologic function as defined by an absolute neutrophil count >= 1,500/mm3, a platelet count >= 100,000/mm3, a WBC >= 3,000/ mm3, and a hemoglobin level of >= 9 g/dl.
* One prior chemotherapy regimen. This may include chemoradiation treatment.
* Disease progression or recurrence within 6 months of last dose of chemotherapy in first chemotherapy regimen.
* At least a 2-week recovery from prior therapy toxicity.
* Signed informed consent.
* Prior CNS involvement by tumor are eligible if previously treated and clinically stable for two weeks after completion of treatment.

Exclusion Criteria:

* Prior Iressa or other EGFR inhibiting agents
* Prior docetaxel therapy
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ.
* Any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy.
* Incomplete healing from previous oncologic or other major surgery.
* Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, St John's Wort, anti-coagulants.
* Absolute neutrophil counts less than 1500 x 109/liter (L) or platelets less than 100,000x 109/liter (L).
* Serum bilirubin greater than 1.25 times the upper limit of reference range (ULRR).
* In the opinion of the investigator, any evidence of severe or uncontrolled systemic disease, (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease).
* A serum creatinine >= 1.5 mg/dl and calculated creatinine clearance <= 60 cc/minute.
* Alanine amino transferase (ALT) or aspartate amino transferase (AST) greater than 2.5 times the ULRR if no demonstrable liver metastases or greater than 5 times the ULRR in the presence of liver metastases.
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial.
* Pregnancy or breast feeding
* The patient has uncontrolled seizure disorder, active neurological disease, or Grade >= 2 neuropathy
* The patient has received any investigational agent(s) within 30 days of study entry.
* The patient has signs and symptoms of keratoconjunctivitis sicca or incompletely treated eye infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-08; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Patient Response Rate to Iressa/Docetaxel | 4 weeks cycles

CONTACTS AND LOCATIONS:
Overall Officials: Edward S. Kim, MD, BS, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org